CLINICAL TRIAL: NCT03568084
Title: Effectiveness of an Intervention in Multicomponent Exercise (MEFAP) in Patients Over 70 Years in Primary Care: Reversibility of Prefrailty
Brief Title: Effectiveness of an Intervention in Multicomponent Exercise in Patients Over 70 Years in Primary Care
Acronym: MEFAP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: SARS-CoV-2 Pandemic
Sponsor: Gerencia de Atención Primaria, Madrid (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PI17/01889
Record Dates: First submitted 2018-05-24; First posted 2018-06-26 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Frail Elderly; Physical Activity
Keywords: elderly; physical activity; exercise; frailty
MeSH Terms: conditions — Motor Activity; Frailty

STUDY DESIGN:
Intervention Model Description: Randomized parallel group multicenter clinical trial. Randomization unit and Unit of analysis: Patient.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MEFAP (Experimental): MEFAP (multicomponent physical activity program) for 12 weekly sessions of an hour and a half which includes 1) briefing 2) exercises for improving aerobic resistance, muscle strength, proprioception-balance and flexibility and 3) delivery of exercise chart to do at home (two times per week).
  Interventions: Other: MEFAP; Other: control usual practice
- Control: usual practice (Active Comparator): No intervention. Individuals allocated to this arm, will be look after as usual in their health Centers.
  Interventions: Other: control usual practice

INTERVENTIONS:
Other: MEFAP — multicomponent physical activity program (MEFAP) with 12 weekly sessions of an hour and a half which includes 1) briefing 2) exercises for improving aerobic resistance, muscle strength, proprioception-balance and flexibility and 3) delivery of exercise chart to do at home (two times per week).
  Arms: MEFAP
Other: control usual practice — Individuals allocated to this arm, will be look after as usual in their health Centers.

SUMMARY:
Objective: To evaluate the effect of a multicomponent physical activity program, compared with the usual medical practice, to reverse prefrailty by Fried in people over 70 years, one year after the end of the intervention.

DETAILED DESCRIPTION:
Objective: To evaluate the effect of a multicomponent physical activity program, compared with the usual medical practice, to reverse prefrailty by Fried in people over 70 years, one year after the end of the intervention.

Location: primary care setting (Madrid Region).

Population: non-dependent and pre-frailty patients ≥ 70 years old, who attend the health centers included in the study.

Design: Randomized parallel group multicenter clinical trial. Randomization unit and Unit of analysis: Patient.

Intervention: multicomponent physical activity program (MEFAP) with 12 weekly sessions of an hour and a half which includes 1) briefing 2) exercises for improving aerobic resistance, muscle strength, proprioception -balance and flexibility and 3) delivery of exercise chart to do at home (two times per week).

Main measures: Main variable: pre-frailty according to Fried phenotype. Secondary variables: sociodemographic, clinical and function variables; adherence, user satisfaction, quality of life.

Analysis: It will be carried out an analysis by intention to treat comparing the retrogression from pre-frailty (1 or 2 Fried criteria) to robust (0 Fried criteria) at the end of the intervention, 6 months after the intervention and one year after the intervention. Cumulative incidence, Relative Risk and Number Needed to Treat with a 95% Confidence Interval. A Generalized Estimating Equation logit model will be adjusted to analyze the associated factors.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged >70 years with a Barthel test ≥90 and pre-frailty (1-2 Fried phenotype frailty criteria).
* For Health Care Centers: Centers who deliver patient to Physiotherapy Units who participate in this Project. Centers where at least two General Practitioners accept to participate in the Project.

Exclusion Criteria:

* Moderate to severe dependency (impairment) for daily living activities (Barthel test <90)
* Enable to achieve Health Care Center for any reason.
* Moderate to severe cognitive impairment (MEC 35 Lobo≤21)
* Severe illness that contraindicates to practice exercise by medical criteria: recent hearth attack (6 months), not controlled arrhythmia, severe hearth valvular disease, not controlled arterial hypertension (systolic blood pressure>180/diastolic blood pressure>100), severe heart failure, severe respiratory failure, diabetes mellitus with frequent acute hypoglycemia, any other circumstance that makes the individual unable to do exercise under medical criteria.

Ages: 70 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 206 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline frail elderly level at one year | one year after the intervention.
  It will be carried out an analysis by intention to treat comparing the retrogression from pre-frailty (1 or 2 Fried criteria) to robust (0 Fried criteria)

SECONDARY OUTCOMES:
Change from baseline frail elderly level at at the end of the intervention (12 weeks) | at the end of the intervention (12 weeks)
  It will be carried out an analysis by intention to treat comparing the retrogression from pre-frailty (1 or 2 Fried criteria) to robust (0 Fried criteria)
Change from baseline frail elderly level at at the at 6 month | 6 month after the intervention
  It will be carried out an analysis by intention to treat comparing the retrogression from pre-frailty (1 or 2 Fried criteria) to robust (0 Fried criteria)
Adherence to intervention | at the end of the intervention (12 weeks)
  degree of adherence to the program (number of sessions with assistance)
Euroqol utilities | at the end of the intervention (12 weeks),
  Euroqol descriptive system (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression)
Visual Analog Scale | at the end of the intervention (12 weeks),
  A Visual Analog Scale with a grade ranging from 0 (the worst possible health status) to 100 (the best possible health status)

CONTACTS AND LOCATIONS:
Locations (1):
- Maria Victoria Castell, Madrid, Spain

REFERENCES:
- [Derived] Castell MV, Gutierrez-Misis A, Sanchez-Martinez M, Prieto MA, Moreno B, Nunez S, Triano R, de Antonio MP, Mateo C, Cano MD, Garrido A, Julian R, Polentinos E, Rodriguez-Barrientos R, Otero Puime A; MEFAP Group. Effectiveness of an intervention in multicomponent exercise in primary care to improve frailty parameters in patients over 70 years of age (MEFAP-project), a randomised clinical trial: rationale and study design. BMC Geriatr. 2019 Jan 28;19(1):25. doi: 10.1186/s12877-018-1024-8. PMID 30691405